CLINICAL TRIAL: NCT03088228
Title: Maternal Periodontal Status and Gingival Crevicular Fluid Levels of Interleukin-6, Interleukin-35, and Interleukin-37 in Preeclampsia
Brief Title: Maternal Periodontal Status and Cytokines in Preeclampsia
Status: Completed | Type: Observational
Sponsor: Hacer Sahin Aydinyurt (Other)
Responsible Party: Sponsor-Investigator, Hacer Sahin Aydinyurt, Principal investigator, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Other Study IDs: 2015-HIZ-DF306
Record Dates: First submitted 2017-02-16; First posted 2017-03-23 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Preeclampsia; Periodontal Diseases
MeSH Terms: conditions — Pre-Eclampsia; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — gingival crevicular flud was analyzed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy pregnants
  Interventions: Diagnostic Test: gingival crevicular fluid collection
- mild preeclampsia
- severe preeclampsia

INTERVENTIONS:
Diagnostic Test: gingival crevicular fluid collection
  Groups: healthy pregnants

SUMMARY:
Background: The purpose of this study is to examine the relationship between maternal preeclampsia and periodontal parameters and the correlation of these two disorders with maternal gingival crevicular fluid levels (GCF) of interleukin (IL)-35, interleukin-37 and interleukin-6. The investigators also investigated their relation to the severity of preeclampsia.

Methods: 82 preeclamptic women were recruited to the study (29 healthy pregnant women, 30 mild preeclamptic patient, 23 severe preeclamptic patient ). The clinical periodontal parameters and GCF samples were collected in the first day of puerperium.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 45 years
* 25 and 40 weeks of gestation.
* Healthy pregnants, mild and severe preeclampsia

Exclusion Criteria:

* Patients with accompanying diseases
* multiple gestations
* congenital abnormalities were excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: 23 severe preeclamptic patient, 30 mild preeclamptic patient and 29 healthy pregnant women were recruited to this study.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
maternal periodontal clinical parameters and IL-37 and IL-35 and IL-6 levels | 6 months
  IL-37 IL-35 and IL-6 levels in maternal gingival crevicular fluid levels between the three groups

IPD SHARING:
Plan to Share IPD: Undecided